CLINICAL TRIAL: NCT04138199
Title: Multi-Center Observational Study to Assess Effectiveness and Safety of Fixed Dose Combination of Generic Product of Lopinavir/Ritonavir in HIV-1 Infected Patients After Switching From Kaletra® (Lopinavir/Ritonavir) for Administrative Reasons in the Routine Clinical Settings of Russian Federation (COPI)
Brief Title: A Study to Assess Effectiveness and Safety of Fixed Dose Combination of Lopinavir/Ritonavir (LPV/r) in Human Immunodeficiency Virus Type 1 (HIV-1) Infected Patients After Switching From Kaletra in the Routine Clinical Settings of Russian Federation
Acronym: COPI
Status: Terminated | Type: Observational
Why Stopped: Strategic Considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-097
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2021-07-06 (Actual); Status verified 2021-07

CONDITIONS: HIV-1 Infection
Keywords: Lopinavir/ritonavir (LPV/r); Kaletra; Human Immunodeficiency Virus (HIV); Generic Product; Highly Active Anti-Retroviral Therapy (HAART)
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Participants with Human Immunodeficiency Virus-1 Infection: Human Immunodeficiency Virus-1 (HIV-1) infected and clinically stable patients on dual or triple HAART including Kaletra who switched or planned to switch to generic product of lopinavir/ritonavir

SUMMARY:
This is a mixed prospective-retrospective, multi-center observational study to assess the virologic effectiveness of generic product of Lopinavir/Ritonavir (LPV/r) after switching from Kaletra in the routine clinical settings of Russian Federation.

ELIGIBILITY:
Inclusion Criteria:

* Human Immunodeficiency Virus Type-1 (HIV-1) infected patients on any dual or triple Highly Active Anti-Retroviral Therapy (HAART) with Kaletra under observation at least 48 weeks and with two consequent plasma HIV-1 RNA levels within the last 24 weeks (plasma HIV-1 RNA level <50 copies/mL) switched to a generic LPV/r as decided by the physician in the routine clinical settings within last 24 weeks from study enrollment date.
* HIV-1 infected patients with last available CD4+ T-cell count test result > 200 cells/mm3 before switching from Kaletra.
* Other (not LPV/r) HAART medicine components of dual or triple HIV therapy not planned to change by regular physician after switching to generic LPV/r.
* Signed Inform Consent form by patient.

Exclusion Criteria:

* Participant has contraindications for the treatment with LPV/r.
* Legal or physical incapability of patient to sign Inform Consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with Human Immunodeficiency Virus Type-1 (HIV-1) infection
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-07-08 (Actual); Study Completion 2020-07-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Who Meet HIV-1- RNA Viral Load >50 Copies/mL, OR CD4+ T-Cell Counts < 200 Cells/mm^3 | Up to 48 Weeks
  Percentage of participants who meet at least one of the following composite endpoint criteria : HIV-1- Ribonucleic Acid (RNA) viral load >50 copies/mL, OR Cluster of differentiation 4 (CD4+) T-cell counts < 200 cells/mm3.
Indicator of Participants Who Have a Development of New or Recurrent Opportunistic Infections or HIV-Associated Malignancies OR any SAE Associated With HIV Treatment | From 48 Weeks Prior to Enrollment through 48 Weeks Post Enrollment
  Percentage of participants who meet at least one of the following composite endpoint criteria: Development of new or recurrent opportunistic infections or HIV-associated malignancies (based on physician observation and decision), OR Any Serious Adverse Event (SAE), associated with HIV treatment.

SECONDARY OUTCOMES:
Time to Failure | Up to Week 48
  Percentage of participants who meet at least one of the following composite endpoint criteria: HIV-1- RNA viral load >50 copies/ml, OR CD4+ T-cell counts < 200 cells/mm3, OR development of new or recurrent opportunistic infections or HIV-associated malignancies (based on physician observation and decision), OR any Serious Adverse Event (SAE), associated with HIV treatment.
Change in HIV-1- RNA Viral Load Compared To The Last Measure On Kaletra Treatment | Up to Week 48
  Untransformed (Absolute) and Base-10 Logarithm Transformed Data Values of HIV-1- RNA Viral Load and The Change As Compared To The Last Measure On Kaletra Treatment
Change in CD4+ T-cell Counts Compared To The Last Measure On Kaletra Treatment | Up to Week 48
  Absolute values of CD4+ T-cell counts the change as compared to the last measure on Kaletra treatment will be summarized with descriptive statistics.
Percentage of Participants With Reasons For Switching From Generic LPV/r To Other Antiretroviral Therapy (ART) For HIV Therapy OR Change In The Dosing Regimen | Up to Week 48
  Percentage of participants with different reasons for switching from generic LPV/r to other products of Antiretroviral Therapy (ART) for HIV therapy or change in the dosing regimen - medical reason (infectiveness, intolerance/toxicity, other), non-medical reasons (lack of availability of generic LPV/r, other) and other reasons.
Percentage of Participants Who Develop HIV Drug Resistance Of Generic LPV/r Treatment | Up to Week 48
  Percentage of participants who develop resistance to each drug will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (10):
- Russia (10):
  - Rep. Cen. of AIDS Profilactis /ID# 216292, Kazan', Tatarstan, Respublika
  - Rep Center for the Prev and Control of AIDS and Inf Dis of the MoH of Chuvashia /ID# 216479, Cheboksary
  - Reg Ctr for AIDS /ID# 216288, Chelyabinsk
  - Reg Ctr for AIDS /ID# 216295, Krasnoyarsk
  - Ctr for AIDS Rostov /ID# 216289, Rostov-on-Don
  - Samara region HIV/AIDS Center /ID# 216290, Samara
  - Mordovian Republican Center for the Prevention and Control of AIDS /ID# 216480, Saransk
  - Saratov Regional Center for the Prevention and Control of AIDS /ID# 216291, Saratov
  - GBUZ Regional Center for the P /ID# 216293, Yekaterinburg
  - GBUZ Sakhalin Regional Center for the Prevention and Control of AIDS /ID# 216478, Yuzhno-Sakhalinsk

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: clinical study report synopsis — https://www.abbvie.com/content/dam/abbvie-dotcom/us/clinical-trials/lopinavir_ritonavir_P20-097.pdf